CLINICAL TRIAL: NCT06977204
Title: Role of Physical Activity on Neuroinflammation in Parkinson's Disease
Brief Title: Physical Activity on Neuroinflammation in Parkinson's Disease
Acronym: MOVE-ON_WP1
Status: Recruiting | Type: Observational
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: MOVE-ON
Record Dates: First submitted 2025-04-28; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Parkinson Disease; Physical Inactivity; Physical Disability
Keywords: Physical activity; Neurological disorder; Neuroinflammation
MeSH Terms: conditions — Parkinson Disease; Sedentary Behavior; Motor Activity; Nervous System Diseases; Neuroinflammatory Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Venous blood samples from the anticubital vein.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- PD-SPORT: In PD-SPORT group the investigators aim to enroll subjects affected by Parkinson's Disease who regularly performed intensive physical activity. For the purpose of this study, the intensive physical activity is defined by the International Physical Activity questionnaire (IPAQ).
- PD-SEDENTARY: In PD-SEDENTARY group the investigators aim to enroll subjects affected by Parkinson's Disease who did not regularly performed intensive physical activity. For the purpose of this study, the intensive of physical activity is defined by the International Physical Activity questionnaire (IPAQ).

SUMMARY:
Parkinson's Disease (PD) is a chronic progressive neurodegenerative disorder clinically defined by the association of resting tremor, rigidity, bradykinesia, and postural instability. The histopathology of PD is characterized by the loss of neurons in the substantia nigra pars compacta (SNPc) and the accumulation of α-synuclein aggregates within Lewy bodies. The pathogenic mechanisms underlying the development of the disease, however, are not yet fully understood: genetics, cellular oxidative stress, mitochondrial dysfunction, environmental factors, and neuroinflammation are all potential mechanisms involved in the pathogenesis of PD.

Several studies have now established the involvement of neuroinflammation in the pathogenesis of PD. It is known that α-synuclein aggregates stimulate microglia and astroglia to secrete pro-inflammatory mediators such as IL 1β, IL6, and TNFα. These molecules activate an inflammatory response characterized by altered blood-brain barrier permeability, leukocyte recruitment, and the expression of other pro-inflammatory cytokines. These events contribute to exposing neurons to oxidative stress and cellular damage. Additionally, cellular damage induces neurons to stimulate the release of DAMPs (Damage Associated Molecular Patterns), which in turn activate glial cells. This creates a state of chronic inflammation that could play a role in the progression of the disease. Supporting this hypothesis, elevated levels of IL1β, IL6, and TNFα have been found in the striatum and SNPc of post-mortem PD samples.

The transcription factor Nrf2 is one of the main regulators of cellular protection in response to stress (inflammation, redox, xenobiotics). Nrf2 promotes the expression of several genes that cooperate in a cytoprotective response, which includes antioxidant defense, resolution of inflammation, increased mitochondrial activity, and protein turnover. Recent clinical studies seem to confirm the hypothesis that Nrf2 plays a role in the pathogenesis of PD, as already suggested by preclinical models. Specifically, altered plasma levels of the Nrf2-activated pathway have been observed in preclinical models.

Studies conducted on animal models of PD have hypothesized how exercise might correlate with protective mechanisms and might promote neuroplasticity and neuro-regeneration, especially when practiced at high intensity. Physical exercise can indeed modulate various systems (including inflammatory pathways and oxidative stress) that regulate neuroinflammation and glial activation. However, the available results are not definitive and often focus on single and separate aspects of the disease.

The aim of the study is to investigate the beneficial effect of physical exercise in patients with Parkinson's Disease (PD). Literature already suggests an improvement in various domains of motor and non-motor aspects, as well as in the overall quality of life, of PD patients even after a period of aerobic activity. Generally, training periods included 3-4 sessions per week of 40-60 minutes each for 4-16 weeks. In general, the literature describes the effects of moderate physical training, while little or nothing is known about how PD is affected by high-intensity sports training.

The primary objective of our study is to compare a group of PD patients undergoing regular and constant intense exercise (PD-sport) with a control group consisting of PD patients leading a sedentary life (PD-sedentary). The primary outcome will be the difference in systemic inflammatory status between the PD-sport group and the PD-sedentary group.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a chronic, progressive neurodegenerative disorder clinically defined by the presence of resting tremor, rigidity, bradykinesia, and postural instability. Pathologically, PD is characterized by the loss of dopaminergic neurons in the substantia nigra pars compacta (SNpc) and the accumulation of α-synuclein aggregates within Lewy bodies. While the precise pathogenic mechanisms underlying PD remain incompletely understood, evidence suggests a multifactorial etiology involving genetic predisposition, oxidative stress, mitochondrial dysfunction, environmental factors, and neuroinflammation.

Emerging research highlights the pivotal role of neuroinflammation in PD pathogenesis. α-Synuclein aggregates are known to activate microglia and astroglia, triggering the release of pro-inflammatory mediators such as IL-1β, IL-6, and TNF-α. This inflammatory response disrupts blood-brain barrier integrity, recruits leukocytes, and amplifies the production of other pro-inflammatory cytokines, exposing neurons to oxidative stress and cellular damage. In turn, neuronal damage promotes the release of damage-associated molecular patterns (DAMPs), perpetuating chronic inflammation. Elevated levels of IL-1β, IL-6, and TNF-α have been detected in the striatum and SNpc of post-mortem PD samples, underscoring the role of inflammation in disease progression.

The transcription factor Nrf2 is a master regulator of cellular defense mechanisms against oxidative and inflammatory stress. Nrf2 orchestrates the expression of genes involved in antioxidant defense, inflammation resolution, mitochondrial activity, and protein turnover. Clinical and preclinical studies suggest that dysregulation of the Nrf2 pathway may contribute to PD pathogenesis, as evidenced by altered plasma levels of Nrf2-regulated pathways in preclinical PD models.

Animal studies have proposed that physical exercise may confer neuroprotective effects by promoting neuroplasticity and neuro-regeneration, particularly through high-intensity training. Exercise has been shown to modulate inflammatory pathways, reduce oxidative stress, and influence glial activation. Despite promising results, most studies have focused on isolated aspects, leaving gaps in our understanding of the comprehensive effects of exercise on PD.

This study aims to investigate the beneficial effects of adapted physical exercise in patients with PD, focusing on its impact on systemic inflammation and secondary outcomes such as gait parameters, functional markers of exercise tolerance, and quality of life.

Study Design

* Observational, case-control, study comparing regular and intense exercise (PD-sport) to a sedentary lifestyle (PD-sedentary).

Primary objective: Evaluate differences in systemic inflammatory status between PD-sport and PD-sedentary groups.

Secondary and Exploratory objective

* Pro- and anti-inflammatory cytokines (IL-6, IL-10, IL-1β, IL-4, IL-17a, TNF-α).
* Plasma extracellular vesicle (EV) profiles (number, size).
* Gait parameters using inertial gait analysis.
* Clinical tests (e.g., MET, 6MWT, UPDRS) and exercise tolerance biomarkers (e.g., VO2peak, gas exchange threshold).
* Psychological outcomes (depression, quality of life, and pain scales).
* Non-motor symptoms (NMS) and cognitive domain assessments.

Recruitment

Participants will be recruited at the IRCCS Mondino Foundation of Pavia, and patient associations. The study will enroll two groups:

1. PD-sport group: Individuals engaging in moderate-to-high-intensity physical activity.
2. PD-sedentary group: Individuals with a sedentary lifestyle. Physical activity levels will be assessed using the short version of the International Physical Activity Questionnaire (IPAQ).

Evaluation

Assessments will include:

Comprehensive clinical evaluation by a movement disorder specialist. Biochemical analysis of inflammatory markers from fasting blood samples (35 mL).

Gait analysis using the G-Walk system. Cognitive and psychological evaluations. Exercise tolerance indices measured via cardiopulmonary exercise testing.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both sexes, aged between 40 and 80 years (extremes included)
* Diagnosis of Parkinson's disease according to the clinical diagnostic criteria of the Movement Disorder Society
* Hoehn & Yahr between 1 and 3

Exclusion Criteria:

* Concomitant diagnosis of other neurological diseases
* Presence of confirmed cognitive decline (MMSE < 24)
* Presence of depression with (BDI > 40)
* Patients with deep brain stimulation implant or undergoing DuoDopa therapy
* Presence of significant diseases affecting the musculoskeletal system
* Presence of internal medicine conditions, considered clinically significant by the investigator
* Acute or recent infections
* Body Mass Index (BMI) >= 30
* Active smoking behavior
* Ongoing treatment with N-acetylcysteine or anti-oxidants
* Pregnancy or lactation

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of individuals diagnosed with Parkinson's disease, but without other clinically relevant medical conditions.
  PD-sport group: this population will include a group of PD subjects who regularly performed a high-intensity and regular physical activity (based on IPAQ questionnaire).
  PD-sedentary group: this population will include a group of PD subjects who did not regularly performed regular physical activity (based on IPAQ questionnaire).
  The absence of other pathological and voluptuary condition is intended to reduce to possible biases of confounders on the inflammatory status.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Set of serum pro-inflammatory and anti-inflammatory cytokines | Single evaluation at baseline
  the investigators will dose a set of of pro-inflammatory and anti-inflammatory cytokines in the serum, namely interleukin 1β (IL-1β), interleukin 2 (IL-2), interleukin 4 (IL-4), interleukin 6 (IL-6), interleukin 10 (IL-10), interleukin 12 (IL-12), tumor necrosis factor alpha (TNF-alpha), and interferon (IFN).

SECONDARY OUTCOMES:
Time Up and Go test | Single evaluation at baseline
  Time Up and Go test (continuous variable with units of measurement: second)
Inertial Gait Analysis | Single evaluation at baseline
  Gait analysis performed Inertial Measeurement Units to assess spatio-temporal variables ( continuous variables: m/s)
Inertial Gait Analysis | Single evaluation at baseline
  Gait analysis performed Inertial Measeurement Units to assess trunk acceleration-derived gait indexes ( continuous variables without measure unit)
5 Sit to Stand Test | Single evaluation at baseline
  Sit to Stand Test (continuous variable with units of measurement: second)
Hand Grip Test | Single evaluation at baseline
  Hand Grip Test (continuous variable with units of measurement: N)
Incremental Maximal Test | Single evaluation at baseline
  Peak oxygen consumption (continuous variable with units of measurement: ml/kg/min)
Geriatric depression scale-30 | Single evaluation at baseline
  Geriatric depression scale-30 (continuous variable, score ranging from 0 to 30 with higher scores indicating more severe depression)
The Parkinson's Disease Questionnaire PDQ-39 | Single evaluation at baseline
  Parkinson's Disease Questionnaire (continuous variable, score ranging from 0 to 156 with higher scores indicating more severe disability)
Brief Pain Inventory (BPI) | Single evaluation at baseline
  Brief Pain Inventory (BPI) (continuous variable, score ranging from 0 to 10 with higher scores indicating more severe disability)
King's PD pain scale (KPPS) | Single evaluation at baseline
  King's PD pain scale (KPPS) (continuous variable, score ranging from 0 to 168 with higher scores indicating more severe pain)
Pain Detect | Single evaluation at baseline
  Pain Detect (continuous variable, score ranging from -1 to 38 with higher scores indicating a more probable neurotic pain)
Peak work rate | Single evaluation at baseline
  Peak work rate (continuous variable with units of measuremente: w)
Peak heart rate | Single evaluation at baseline
  Peak heart rate (continuous variable with units of measuremente: b/min)
Gas exchange threshold | Single evaluation at baseline
  Gas exchange threshold (continuous variable with units of measuremente: l/min)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Mondino Foundation, Pavia, Pavia, Italy

REFERENCES:
- [Background] Szymura J, Kubica J, Wiecek M, Pera J. The Immunomodulary Effects of Systematic Exercise in Older Adults and People with Parkinson's Disease. J Clin Med. 2020 Jan 9;9(1):184. doi: 10.3390/jcm9010184. PMID 31936624
- [Background] Xu J, He X, Xu Y, Chen X, Li M, Zhang L, Fu X, Pan M, Wang Q, Hu X. Characteristics of systemic inflammation and brain iron deposition in Parkinson's disease patients. Ann Clin Transl Neurol. 2022 Mar;9(3):276-285. doi: 10.1002/acn3.51512. Epub 2022 Jan 25. PMID 35078271
- [Background] Pajares M, I Rojo A, Manda G, Bosca L, Cuadrado A. Inflammation in Parkinson's Disease: Mechanisms and Therapeutic Implications. Cells. 2020 Jul 14;9(7):1687. doi: 10.3390/cells9071687. PMID 32674367